CLINICAL TRIAL: NCT02913651
Title: Cardiovascular Variability and Heart Rate Arousal Response in Idiopathic Hypersomnia
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1600111
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-09

CONDITIONS: Narcolepsy; Cataplexy
Keywords: Idiopathic hypersomnia; heart rate variability; parasympathetic activity; autonomic arousal response
MeSH Terms: conditions — Narcolepsy; Cataplexy; Idiopathic Hypersomnia | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic hypersomnia: Drug-free patients diagnosed with idiopathic hypersomnia from 01/01/11 to 15/09/15
  Interventions: Device: Polysomnography
- Controls: Patients with no sleep complaints, having a 24-h ambulatory ad libitum polysomnography
  Interventions: Device: Polysomnography

INTERVENTIONS:
Device: Polysomnography — The polysomnography, for both groups, was performed accordance with standard practice

SUMMARY:
Autonomic nervous system dysfunction has been described in narcolepsy with cataplexy affecting the sympathetic function. In this study the investigators analyzed whether altered diurnal and nocturnal cardiovascular control is present in idiopathic hypersomnia. Drug-free patients diagnosed with idiopathic hypersomnia and age-matched controls were included. Clinical data, 24-h polysomnography, heart rate variability and the heart rate response to spontaneous arousal are analyzed.

ELIGIBILITY:
Inclusion Criteria:

Idiopathic hypersomnia patients

* idiopathic hypersomnia diagnosis
* complaints of excessive daytime sleepiness for >1 year
* a night-time length >10 h for 3 weeks before polysomnography as assessed by a sleep diary

Inclusion Criteria:

no idiopathic hypersomnia patients

* no sleep complaints and excessive daytime sleepiness (Epworth sleep questionnaire score <10

Exclusion Criteria (both):

* Narcolepsy-cataplexy
* sleep irregularities and sleep deprivation symptoms
* lack of neurological or psychiatric diseases
* upper airway resistance syndrome
* periodic limbs movements
* cerebral lesion
* medication or drinks affecting sleep and wake state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic hypersomnia patients and no idiopathic hypersomnia patient
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
High Frequencies (HF) | During the polysomnography (one night)
  Nocturnal parasympathetic activity (HF parameter of heart rate variability analysis)

SECONDARY OUTCOMES:
Heart rate variability (HRV) | During the polysomnography (one night)
  HRV is measured by the polysomnography. It is a composite outcome : Standard Deviation of NN intervals (SDNN), the proportion of NN30 (and 50) divided by total number of NNs (pNN30, pNN50), Root Mean Square of Successive Differences (RMSSD), Standard Deviation type 1 and 2 (SD1, SD2), Low Frequencies (LF), Very Low Frequencies (VLF), LF/HF ratio and Ptot indexes
Apnea-Hypopnea Index (AIH) | During the polysomnography (one night)
Epworth Sleepiness Scale (ESS) | Before the polysomnography (one night)
  It examines eight different situations using a 4-grade scale ranging from 0 (no chances of napping) to 3 (high chances of napping). Subjects were defined as sleepy if they had an ESS>10

CONTACTS AND LOCATIONS:
Overall Officials: Emilia SFORZA, MD, Study Chair — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No